CLINICAL TRIAL: NCT00162422
Title: The Effect of β2 Genetic Polymorphisms on the Brochodilatation Effect of Albuterol ex-Vivo
Brief Title: Genetic Determinants of the Bronchodilatation Effect of Albuterol ex-Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yc19557-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

INTERVENTIONS:
Drug: albuterol

SUMMARY:
The role played by ß2AR polymorphisms in determining the bronchial response to ß2AR agonist drugs, has been confirmed by several studies.

The purpose of the present study is to examine possible causal relationships between genetically based alteration in the structure of ß2AR and drug responsiveness. An ex-vivo model (organ bath technique) will be used to investigate association between polymorphisms in the coding region of ß2AR and the response of bronchial rings derived from human lung tissue to the respective agonists (i.e. salbutamol).

In the second part of the study the same bronchial rings will be incubated for 24 hours in a solution containing fixed concentration of albuterol. A second dose response curve for rising concentrations of albuterol will be constructed and a relationship between β2 genetic polymorphisms and the extent of desensitization to albuterol will be investigated.

In addition, through specifically designed receptor binding assay the bronchial tissue will be used to define the affinity (Kd) and expression (Vmax) of the ß2 receptor. These data will enable to enhance our understanding regarding the mechanism responsible for the association noted between ß2AR polymorphism and altered drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Macroscopically normal pulmonary tissue

Exclusion Criteria:

* The presence of pathological finding in the pulmonary tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-08

PRIMARY OUTCOMES:
The extent of bronchial dilatation ex-vivo
The extent of decrease in brochial dilatation after prolonged incubation with albuterol

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, ND, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel